CLINICAL TRIAL: NCT06007911
Title: Venetoclax-Navitoclax With Cladribine-based Salvage Therapy in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor withdrew support.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Guru Subramanian Guru Murthy, Assistant Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00050186
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Relapsed Adult AML; Refractory AML
Keywords: Acute Myeloid Leukemia; AML; Venetoclax; Navitoclax; cladribine-based salvage therapy; CLAG-M
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — navitoclax; venetoclax; Cladribine; Cytarabine; Mitoxantrone; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cladribine-Low Dose Cytarabine Backbone Dose Level -1 (Experimental): Dose level -1 will be considered only if there are dose-limiting toxicities at dose level 0. This is a regimen of navitoclax, venetoclax, cladribine and cytarabine.
  Interventions: Drug: Navitoclax Dose Level -1; Drug: Venetoclax Dose Level -1; Drug: Cladribine; Drug: Cytarabine (Cladribine Low Dose Cytarabine Backbone)
- Cladribine-Low Dose Cytarabine Backbone Dose Level 0 (Experimental): This is a regimen of navitoclax, venetoclax, cladribine and cytarabine.
  Interventions: Drug: Navitoclax Dose Level 0; Drug: Venetoclax Dose Levels 0 to 2; Drug: Cladribine; Drug: Cytarabine (Cladribine Low Dose Cytarabine Backbone)
- Cladribine-Low Dose Cytarabine Backbone Dose Level 1 (Experimental): This is a regimen of navitoclax, venetoclax, cladribine and cytarabine.
  Interventions: Drug: Navitoclax Dose Level 1; Drug: Venetoclax Dose Levels 0 to 2; Drug: Cladribine; Drug: Cytarabine (Cladribine Low Dose Cytarabine Backbone)
- Cladribine-Low Dose Cytarabine Backbone Dose Level 2 (Experimental): This is a regimen of navitoclax, venetoclax, cladribine and cytarabine.
  Interventions: Drug: Navitoclax Dose Level 2; Drug: Venetoclax Dose Levels 0 to 2; Drug: Cladribine; Drug: Cytarabine (Cladribine Low Dose Cytarabine Backbone)
- Cladribine-Low Dose Cytarabine Backbone Dose Maximum Tolerated Dose (MTD) (Experimental): The MTD is the highest dose level at which no more than 1 of 6 treated participants, experiences a dose-limiting toxicity.
  Interventions: Drug: Navitoclax Dose Level -1; Drug: Navitoclax Dose Level 0; Drug: Navitoclax Dose Level 1; Drug: Navitoclax Dose Level 2; Drug: Venetoclax Dose Level -1; Drug: Venetoclax Dose Levels 0 to 2; Drug: Cladribine; Drug: Cytarabine (Cladribine Low Dose Cytarabine Backbone)
- CLAG-M Backbone Level -1 (Experimental): Dose level -1 will be considered only if there are dose-limiting toxicities at dose level 0. This is a regimen of navitoclax, venetoclax, cladribine, cytarabine, mitoxantrone and G-CSF.
  Interventions: Drug: Navitoclax Dose Level -1; Drug: Venetoclax Dose Level -1; Drug: Cladribine; Drug: Cytarabine (CLAG-M Backbone); Drug: Mitoxantrone; Drug: Granulocyte Colony-Stimulating Factor
- CLAG-M Backbone Level 0 (Experimental): This is a regimen of navitoclax, venetoclax, cladribine, cytarabine, mitoxantrone and granulocyte colony-stimulating factor (G-CSF).
  Interventions: Drug: Navitoclax Dose Level 0; Drug: Venetoclax Dose Levels 0 to 2; Drug: Cladribine; Drug: Cytarabine (CLAG-M Backbone); Drug: Mitoxantrone; Drug: Granulocyte Colony-Stimulating Factor
- CLAG-M Backbone Level 1 (Experimental): This is a regimen of navitoclax, venetoclax, cladribine, cytarabine, mitoxantrone and G-CSF.
  Interventions: Drug: Navitoclax Dose Level 1; Drug: Venetoclax Dose Levels 0 to 2; Drug: Cladribine; Drug: Cytarabine (CLAG-M Backbone); Drug: Mitoxantrone; Drug: Granulocyte Colony-Stimulating Factor
- CLAG-M Backbone Level 2 (Experimental): This is a regimen of navitoclax, venetoclax, cladribine, cytarabine, mitoxantrone and G-CSF.
  Interventions: Drug: Navitoclax Dose Level 2; Drug: Venetoclax Dose Levels 0 to 2; Drug: Cladribine; Drug: Cytarabine (CLAG-M Backbone); Drug: Mitoxantrone; Drug: Granulocyte Colony-Stimulating Factor
- CLAG-M Backbone Maximum Tolerated Dose (Experimental): The MTD is the highest dose level at which no more than 1 of 6 treated participants, experiences a dose-limiting toxicity.
  Interventions: Drug: Navitoclax Dose Level -1; Drug: Navitoclax Dose Level 0; Drug: Navitoclax Dose Level 1; Drug: Navitoclax Dose Level 2; Drug: Venetoclax Dose Level -1; Drug: Venetoclax Dose Levels 0 to 2; Drug: Cladribine; Drug: Cytarabine (CLAG-M Backbone); Drug: Mitoxantrone; Drug: Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: Navitoclax Dose Level -1 — 25 mg by mouth on days 1-7.
  Other Names: ABT-263
  Arms: CLAG-M Backbone Level -1; CLAG-M Backbone Maximum Tolerated Dose; Cladribine-Low Dose Cytarabine Backbone Dose Level -1; Cladribine-Low Dose Cytarabine Backbone Dose Maximum Tolerated Dose (MTD)
Drug: Navitoclax Dose Level 0 — 50 mg by mouth on days 1-10.
  Other Names: ABT-263
  Arms: CLAG-M Backbone Level 0; CLAG-M Backbone Maximum Tolerated Dose; Cladribine-Low Dose Cytarabine Backbone Dose Level 0; Cladribine-Low Dose Cytarabine Backbone Dose Maximum Tolerated Dose (MTD)
Drug: Navitoclax Dose Level 1 — 75 mg by mouth on days 1-10.
  Other Names: ABT-263
  Arms: CLAG-M Backbone Level 1; CLAG-M Backbone Maximum Tolerated Dose; Cladribine-Low Dose Cytarabine Backbone Dose Level 1; Cladribine-Low Dose Cytarabine Backbone Dose Maximum Tolerated Dose (MTD)
Drug: Navitoclax Dose Level 2 — 100 mg by mouth on days 1-10.
  Other Names: ABT-263
  Arms: CLAG-M Backbone Level 2; CLAG-M Backbone Maximum Tolerated Dose; Cladribine-Low Dose Cytarabine Backbone Dose Level 2; Cladribine-Low Dose Cytarabine Backbone Dose Maximum Tolerated Dose (MTD)
Drug: Venetoclax Dose Level -1 — 400 mg by mouth on days 1-7.
  Other Names: Venclexta
  Arms: CLAG-M Backbone Level -1; CLAG-M Backbone Maximum Tolerated Dose; Cladribine-Low Dose Cytarabine Backbone Dose Level -1; Cladribine-Low Dose Cytarabine Backbone Dose Maximum Tolerated Dose (MTD)
Drug: Venetoclax Dose Levels 0 to 2 — 400 mg by mouth on days 1-14.
  Other Names: Venclexta
  Arms: CLAG-M Backbone Level 0; CLAG-M Backbone Level 1; CLAG-M Backbone Level 2; CLAG-M Backbone Maximum Tolerated Dose; Cladribine-Low Dose Cytarabine Backbone Dose Level 0; Cladribine-Low Dose Cytarabine Backbone Dose Level 1; Cladribine-Low Dose Cytarabine Backbone Dose Level 2; Cladribine-Low Dose Cytarabine Backbone Dose Maximum Tolerated Dose (MTD)
Drug: Cladribine — 5 mg/m^2 intravenously days 1-5.
  Other Names: Mavenclad; Leustatin DSC
Drug: Cytarabine (Cladribine Low Dose Cytarabine Backbone) — 20 mg/m^2 subcutaneous days 1-10.
  Other Names: ara-C
  Arms: Cladribine-Low Dose Cytarabine Backbone Dose Level -1; Cladribine-Low Dose Cytarabine Backbone Dose Level 0; Cladribine-Low Dose Cytarabine Backbone Dose Level 1; Cladribine-Low Dose Cytarabine Backbone Dose Level 2; Cladribine-Low Dose Cytarabine Backbone Dose Maximum Tolerated Dose (MTD)
Drug: Cytarabine (CLAG-M Backbone) — 1.5 g/m^2 intravenously days 1-5.
  Other Names: ara-C
  Arms: CLAG-M Backbone Level -1; CLAG-M Backbone Level 0; CLAG-M Backbone Level 1; CLAG-M Backbone Level 2; CLAG-M Backbone Maximum Tolerated Dose
Drug: Mitoxantrone — 10 mg/m^2 intravenously days 1-3.
  Other Names: Novantrone
  Arms: CLAG-M Backbone Level -1; CLAG-M Backbone Level 0; CLAG-M Backbone Level 1; CLAG-M Backbone Level 2; CLAG-M Backbone Maximum Tolerated Dose
Drug: Granulocyte Colony-Stimulating Factor — 300 mcg subcutaneously days 1-5.
  Other Names: G-CSF; filgrastim; Neupogen
  Arms: CLAG-M Backbone Level -1; CLAG-M Backbone Level 0; CLAG-M Backbone Level 1; CLAG-M Backbone Level 2; CLAG-M Backbone Maximum Tolerated Dose

SUMMARY:
This is an open-label phase I study designed to evaluate the safety of venetoclax-navitoclax with cladribine-based salvage therapy.

DETAILED DESCRIPTION:
The primary objective of the study is to determine a maximum-tolerated dose (MTD) combination of venetoclax-navitoclax with cladribine-based salvage therapy. Subjects will be entered sequentially to each dose level. For each dose level, if none of the first three subjects at that level experiences a dose-limiting toxicity (DLT), new subjects may be entered at the next higher dose level. If one of three subjects experience a DLT, up to three more subjects are to be treated at that same dose level. If none of the additional three subjects at that dose level experiences a DLT, new subjects may be entered at the next higher dose level. However, if one or more of the additional three subjects experience a DLT, then no further subjects are to be started at that dose level and either de-escalate one level or if the preceding dose is already completed then that dose is the MTD. The MTD will be defined as the highest dose level at which none of the first three treated subjects, or no more than one of the first six treated subjects, experiences a DLT.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years or older.
2. Patients must have a diagnosis of morphologically documented AML or secondary AML from prior conditions, such as myelodysplastic syndrome (MDS), myeloproliferative neoplasm (MPN), MDS/MPN, chronic myelomonocytic leukemia (CMML) or therapy-related AML (t-AML), as defined by the World Health Organization (WHO) 2022 criteria.
3. Relapsed or refractory to at least one prior line of therapy.
4. Previous therapy with venetoclax.
5. Eastern Cooperative Oncology Group (ECOG) performance status of:

   1. 0-3 for Arm A (i.e., Cladribine-low dose cytarabine backbone arm).
   2. 0-2 for Arm B (i.e., CLAG-M backbone arm).
6. Left ventricular ejection fraction (LVEF) of:

   1. LVEF ≥35% for Arm A (i.e., Cladribine-low dose cytarabine backbone arm).
   2. LVEF ≥45% for Arm B (i.e., CLAG-M backbone arm).
7. Creatinine clearance (CrCl) as calculated by the Cockroft-Gault formula, of:

   1. CrCl ≥ 30 mL/min for Arm A (i.e., Cladribine-low dose cytarabine backbone arm).
   2. CrCl ≥ 40 mL/min for Arm B (i.e., CLAG-M backbone arm).
8. Clinical laboratory values within the following parameters:

   1. Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN) unless attributable to underlying leukemia. Patient with total bilirubin > 1.5 × institutional ULN may enroll if direct bilirubin ≤ 1.5 × institutional ULN of the direct bilirubin.
   2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × institutional ULN, unless attributable to underlying leukemia.
   3. White blood cell (WBC) count < 25,000/µL before Cycle 1, Day 1 of therapy (Note: Hydroxyurea, cytarabine or leukapheresis may be used to meet this criterion.)
   4. Platelet count of at least 20,000/µL before Cycle 1, Day 1 of therapy (Note: Platelet transfusion can be used to meet this criterion.)
9. Female subjects who:

   1. Are postmenopausal for at least one year before the screening visit, OR
   2. Are surgically sterile, OR
   3. If they are of childbearing potential:

   i. Agree to practice one highly effective method and one additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through four months after the last dose of study drug (female and male condoms should not be used together), OR ii. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception).
10. Male subjects, even if surgically sterilized (i.e., status post vasectomy), who:

    1. Agree to practice effective barrier contraception during the entire study treatment period from the time of signing the informed consent through and through four months after the last dose of study drug (female and male condoms should not be used together), OR
    2. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)
11. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Acute promyelocytic leukemia.
2. Prior therapy with B-cell lymphoma-extra large (BCL-XL) inhibitor.
3. Treatment with systemic antineoplastic therapy within 14 days or five half-lives from the last dose - whichever is longer - before Cycle 1, Day 1 of therapy. Radiation within 14 days before Cycle 1, Day 1 of therapy. The use of hydroxyurea/cytarabine for leukoreduction is permitted.
4. Hematopoietic stem cell transplantation (HCT) or chimeric antigen receptor T-cell therapy (CAR-T cell) within 60 days of enrollment. (If patients had prior allogeneic HCT, they should have no active graft-versus-host disease and should be off calcineurin inhibitors at least four weeks prior to cycle 1 day 1 of therapy.)
5. Current systemic treatment with strong or moderate Cytochrome P4503A (CYP3A) inducers within 7 days prior to Cycle 1, Day 1 of therapy.
6. Presence of another active malignancy requiring systemic treatment within the last 12 months, except for localized cancers that have been adequately treated.
7. Known HIV positive patients who DO NOT meet the following criteria:

   1. Cluster of differentiation (CD) 4 count > 350 cells/mm^3.
   2. Undetectable viral load.
   3. Maintained on modern therapeutic regimens utilizing non-CYP-interactive agents.
   4. No history of AIDS-defining opportunistic infections.
8. Known hepatitis B surface antigen seropositive or active hepatitis C infection. Note: Patients who have isolated positive hepatitis B core antibody (i.e., in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load. Patients who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load.
9. Female subjects who are both lactating and breastfeeding or of childbearing potential who have a positive serum test during screening.
10. Female subjects who intend to donate eggs (ova) during the course of the study or four months after receiving their last dose of the study drug(s).
11. Male subjects who intend to donate sperm during the course of this study or four months after receiving their last dose of the study drug(s).
12. Has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or star fruit from three days prior to Cycle 1, Day 1 to throughout the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-31 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose of Navitoclax for the Cladribine-Low Dose Cytarabine Backbone | Up to three years
  The dose identified in this trial that will be used in future clinical trials.
Recommended Phase 2 Dose for Navitoclax for the CLAG-M Backbone | Up to three years
  The dose identified in this trial that will be used in future clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Guru Subramanian Guru Murthy, MD, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No